CLINICAL TRIAL: NCT06932120
Title: Technology-supported Interventions for Prolonged Grief Disorder in Adults a Randomized Controlled Trial
Brief Title: Technology-supported Interventions for Prolonged Grief Disorder (PGD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UJaumeI_iGROw_1
Record Dates: First submitted 2025-03-17; First posted 2025-04-17 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Prolonged Grief Disorder (PGD)
Keywords: Prolonged grief disorder; Efficacy; Randomized controlled trial; Internet-based treatment; blended intervention; Ecological Momentary Assessment (EMA); Ecological Momentary Intervention (EMI)
MeSH Terms: conditions — Prolonged Grief Disorder

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial with two treatment conditions and one WL control condition: a three-armed simple-blind RCT. Patients will be assessed for eligibility and if they meet the inclusion criteria, they will be randomly allocated to one of the three experimental conditions (BF-Grow, iGROw and WL group). The allocation schedule will be generated through an independent researcher who will be unaware of the characteristics of the study. Patients will agree to participate before the random allocation and without knowing to which treatment they will be assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BF-Grow group: Blended Format group (Experimental): Arm 1: Experimental. BF-Grow group. Patients of the BF-GROw group will receive a treatment module every 10-12 days, in addition to an individual session by videoconference (approximately 30 minutes). In total they will receive between 8-10 sessions with the therapist. During these sessions, the therapist will be resolved.
  Interventions: Behavioral: Internet-based treatment (GROw) combined with face-to-face videoconferencing sessions with a therapist in BF-GROw group
- iGROw group: Self-applied online format group (Experimental): Arm 2: Experimental. iGrow group. Patients of the iGrow group will carry out the treatment in a totally self-applied way. They will be able to access the next module once 7 days have elapsed since the start of the previous one. The total time of access to treatment will be about 12-14 weeks. This condition will be supported by the App developed which contains the EMA and EMI tools.
  Interventions: Behavioral: Internet-based treatment (GROw) supported by the App developed which contains the EMA and EMI tools in iGROw group.
- Waiting List (WL) control group (No Intervention): Arm 3: Waiting List control group. Participants in the WL will answer the pre- and post-evaluation and they will be randomly assigned to one of the two treatment conditions after spending time on the waiting list (10-12 weeks) for ethical reasons.

INTERVENTIONS:
Behavioral: Internet-based treatment (GROw) combined with face-to-face videoconferencing sessions with a therapist in BF-GROw group — The treatment that will be applied is an internet-based treatment (GROw) (Tur et al., 2021, 2022)combined with face-to-face videoconferencing sessions with a therapist (blended) . This protocol has 8 weekly modules and lasts between 8 and 12 weeks. The modules included are: 1) Welcome (starting the program), 2) Understanding reactions to loss, 3) Coping with loss, 4) Loss integration and restoration (first steps), 5) Deeping integration and restoration of loss, 6) Consolidating loss integration and restoration, 7) Self-care, guilt, and forgiveness in the grieving process, and 8) Evaluating progress and looking to the future. BF-GROw group will receive a treatment module every 10-12 days. This protocol is available online: (https://psicologiaytecnologia.labpsitec.es).
  Arms: BF-Grow group: Blended Format group
Behavioral: Internet-based treatment (GROw) supported by the App developed which contains the EMA and EMI tools in iGROw group. — The treatment that will be applied is an internet-based treatment (GROw) (Tur et al., 2021, 2022) supported by the App developed which contains the Ecological Momentary Assessment (EMA) and Ecological Momentary Intervention (EMI) tools . This protocol has 8 weekly modules and lasts between 8 and 12 weeks. The modules included are: 1) Welcome (starting the program), 2) Understanding reactions to loss, 3) Coping with loss, 4) Loss integration and restoration (first steps), 5) Deeping integration and restoration of loss, 6) Consolidating loss integration and restoration, 7) Self-care, guilt, and forgiveness in the grieving process, and 8) Evaluating progress and looking to the future. This protocol is available online: (https://psicologiaytecnologia.labpsitec.es).
  Arms: iGROw group: Self-applied online format group

SUMMARY:
The main aim of this project is to test the efficacy of two formats of delivering an internet- based treatment(GROw) for Prolonged Grief Disorder (PGD) in order to enhance treatment adherence: in a blended format (that combines self-applied treatment online with face-to face sessions with a therapist by videoconference: BF-GROw) and self-applied online format supported by Ecological Momentary Assessment (EMAs) and Ecological Momentary Interventions (EMIs) (iGROw), compared with a waiting list (WL) control group in a community sample of patients with the diagnosis of PGD. The general initial hypothesis is that both treatment conditions (blended format and self-applied format supported by EMAs and EMIs) will significantly produce an improvement in grief symptoms, compared to the WL control group.

DETAILED DESCRIPTION:
The grieving process is defined as a painful response, including cognitive, emotional and behavioural components, following the death of a loved one. This response of unique intensity and duration for each individual may involve symptoms such as intense emotions, worry, memories of the deceased and a decrease in activity, which will diminish over time. However, it is estimated that 10% of the population who experience the death of a loved one eventually develop prolonged grief disorder (PGD). There are now evidence-based psychological treatments that are effective in treating PGD. However, 70% of people who need them do not receive them. According to the scientific literature, self-administered technology-supported interventions have been developed to treat this problem and have demonstrated multiple benefits. This study aims to test the efficacy and efficiency of different treatment options that exist for this disorder through a randomized controlled trial. Participants will be adults with a diagnosis of PGD, according to ICD-11 criteria for PGD (WHO,2018) and will be randomly distributed into three groups: 1) blended intervention (BF-Grow group); 2) self-applied intervention supported by EMAs and EMIs (iGrow group); and 3) waiting-list group (WL control group). Both treatment groups will receive the same treatment (GROw) consisting of 8 modules: 1. Welcoming, 2. Understanding reactions to loss, 3. Coping with loss, 4. Loss integration and restoration (first steps), 5. Deepening integration and restoration of loss, 6. Consolidating loss integration and restoration, 7. Self-care, guilt and forgiveness in the grieving process and 8. Evaluating progress and looking to the future.

On the one hand, group 1 (BF-Grow) will receive a treatment module every 10-12 days and in addition an individual session of approximately 30 minutes with a therapist. On the other hand, group 2 (iGrow) will carry out the entire intervention on a self-applied basis only and will be able to access the next module 7 days after the start of the previous one. In addition, this condition will be supported by an App which contains EMA and EMI tools. Participants will be evaluated at baseline, post-treatment, and 3- and 12-month follow-ups.

This study will follow the Consolidated Standards for Reporting Trials (CONSORT)statement and the SPIRIT guidelines (Standard Protocol Items: Recommendations for Intervention Trials).

Specific objectives of the study include: examine the efficacy of BF-Grow and iGROw intervention formats compared to a WL group in the post-treatment and In addition, post hoc comparisons will be conducted among the adjusted means of the three groups.

ELIGIBILITY:
Inclusion Criteria:

* Being at least 18 years old.
* Meeting diagnostic criteria for Prolonged Grieft Disorder based on the International Classification of Diseases 11 edition (ICD-11).
* Sign an informed consent.
* Ability to understand and read Spanish.
* Ability to use a computer.
* Having an e-mail address.
* Having an internet connection and Access to a Smartphone.

Exclusion Criteria:

* Presence of high risk of suicide.
* Presence of axis I severe mental disorder: substance abuse or dependence, psychotic disorder, dementia, bipolar disorder; severe personality disorder or medical illness whose severity or characteristics prevent treatment.
* Receiving other psychological treatment during the study.
* An increase and/or change in the medication during the study period, in the case of receiving pharmacological treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2026-11-10 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in the Inventory of Complicated Grief (ICG). | Immediately prior to treatment, Immediately after treatment, 3 months after treatment, 12 months after treatment
  The Inventory of Complicated Grief (ICG) is a self-administered instrument that assesses grief symptoms in adults. It is a simple instrument that allows distinguishing normal grief reactions from complicated ones.The instrument consists of 19 items written in the first person with five response options (Likert): 0; never 1; rarely 2; sometimes 3; often and 4; always. about the client's thoughts and behaviors related to immediate grief. The items assess the frequency of emotional, cognitive and behavioral symptoms characteristic of the grieving process.

SECONDARY OUTCOMES:
Change in Beck Depression Inventory-II (BDI-II). | Immediately prior to treatment, immediately after treatment, 3 months after treatment, 12 months after treatment.
  It is a self-report measure composed of 21 items that assess the severity of depressive symptomatology in the last two weeks. It uses a response scale from 0 to 3, with higher scores indicating greater severity. It is calculated by adding the score of the 21 items and the maximum total score is 63.
Change in Typical Beliefs Questionnaire (TBQ). | Immediately prior to treatment, immediately after treatment, 3 months after treatment, 12 months after treatment.
  A 25-item self-report instrument that assesses cognitions that hinder adjustment to loss. Structured in five factors: "Protesting the death", "Negative thoughts about the world", "Needing the person", "Less grief is a mistake" and "Suffering too much". It measures the degree of agreement regarding different affirmations using a Likert-type response system ranging from 0 (not at all) to 4 (strongly agree). A total score from 0 to 100 is calculated by adding up all the items.
Change in Overall Anxiety Severity and Impairment Scale (OASIS). | Immediately prior to treatment, immediately after treatment, 3 months after treatment, 12 months after treatment.
  It is a self-applied instrument that assesses the frequency and severity of anxiety symptoms. It also measures the degree of avoidance and interference in all areas of the patient's life. It consists of 5 items with a response scale from 0 to 4. Higher scores indicate greater severity or frequency of symptomatology. The maximum score is 20 and is calculated by adding the score obtained for each of the 5 items.
Change in Overall Depression Severity and Impairment Scale (ODSIS). | Immediately prior to treatment, immediately after treatment, 3 months after treatment, 12 months after treatment.
  It is a self-applied instrument that assesses the frequency and severity of depression symptoms. It also measures the degree of avoidance and interference in all areas of the patient's life. It consists of 5 items with a response scale from 0 to 4. One additional item has been included to assess suicide ideation. The maximum score is 20 and is calculated by adding the score obtained for each of the 5 items.
Change in Short-Form of the International Positive and Negative Affect Schedule (iPANAS). | Immediately prior to treatment, immediately after treatment, 3 months after treatment, 12 months after treatment.
  The International Positive and Negative Affect Schedule Short Form (I-PANAS-SF) is a shortened version of the original 20-item PANAS to measure two dimensions of affect, positive and negative affect. The scale is composed of 10 items using a Likert-type scale with assigned scores of: Not at all (0); A little (1); Quite a lot (2); A lot (3); Very much (4). The person rates a list of words describing feelings and emotions that people have, indicating to what extent they describe how he/she has been feeling lately.

OTHER OUTCOMES:
Change in Structured Clinical Interview for Complicated Grief (SCI-CG). | Immediately prior to treatment, immediately after treatment, 3 months after treatment, 12 months after treatment.
  The SCI-CG is a 31-item clinician-administered instrument to assess the presence of complicated grief symptoms. Each item is answered on a 3-point Likert-type scale (Not present, Unsure or misleading, and Present). The maximum score is 93 and is calculated by adding the scores for each item.
Change in Anxiety Disorders Interview Schedule (ADIS) Clinician Severity rating Scale . | Immediately prior to treatment, immediately after treatment, 3 months after treatment, 12 months after treatment.
  This instrument assesses the severity of symptoms evaluated by the clinician and the scale ranged from 0-8.Clinicians assign ratings from 0 (absent) to 8 (very severely disabling) reflecting the intensity of symptoms, associated avoidance, and interference with functioning. Higher scores indicating greater severity.
Change in Quality of Life Index (QLI). | Immediately prior to treatment, immediately after treatment, 3 months after treatment, 12 months after treatment.
  It is a self-administered instrument that includes 10 items that evaluate the patients' quality of life in different areas and in a global manner. It uses a 10-point Likert-type scale: 1 (poor) to 10 (excellent).Higher scores indicate improvement.
Change in The Work and Social Adjustment Scale (WSAS). | Immediately prior to treatment, immediately after treatment, 3 months after treatment, 12 months after treatment.
  It is a self-administered instrument that assesses psychosocial functional impairment. It consists of 5 items that are scored on a scale from 0 (not at all) to 8 (very severe). The maximum score is 40 and is calculated by adding the score of all items, the higher the score, the greater the interference in different areas.
Change in Posttraumatic Growth Inventory (PTGI). | Immediately prior to treatment, immediately after treatment, 3 months after treatment, 12 months after treatment.
  It is a self-administered instrument consisting of 21 items that assess growth and coping after having experienced an adverse or traumatic event. It uses a likert scale ranging from 0 (I did not experience this change as a consequence of the crisis) to 5 (I experienced this change to a great extent), with a higher score indicating a greater positive transformation.
Change in The Purpose-In-Life Test (PIL- 10). | Immediately prior to treatment, Immediately after treatment, 3 months after treatment, 12 months after treatment
  It is a self-administered instrument consisting of 10 questions that evaluates different aspects of the meaning of life. It uses a response scale from 1 to 7. Higher scores indicate a greater sense of life and the maximum score is 70.
Change in The Five-Facet Mindfulness Questionnaire (FFMQ-15). | Immediately prior to treatment, Immediately after treatment, 3 months after treatment, 12 months after treatment
  It evaluates five facets of mindfulness (Observing, Describing, Acting with awareness, Non judging internal experience, Non reactivity to internal experience). It consists of 15 items that are answered on a 5-point Likert scale ranging from 1 ("never or very rarely true") to 5 ("very often or always true"). Higher scores represent higher dispositional mindfulness. It shows good internal consistency in the 5 scales.
Change in The Self-Compassion Scale-Short Form (SCS-SF). | Immediately prior to treatment, Immediately after treatment, 3 months after treatment, 12 months after treatment
  It is a 12-item self-administered instrument that assesses the capacity for self-compassion. To calculate the total self-compassion score, a total mean is calculated taking into account the inverse items. The subscale scores are calculated by calculating the mean of the responses of the subscale items.
Scale of expectation and satisfaction with the treatment. | Scale of expectation: Immediately prior to treatment. Scale of satisfaction: Immediately after treatment.
  These two scales consist of six items each. Participants rate these items on a scale from 0 (strongly disagree) to 10 (strongly agree). Their aim is to evaluate the treatment's ability to meet the patients' expectations, its perceived logic, its potential for treating other psychological issues, its usefulness for the patient, the likelihood of recommending it to others and its aversion. The Expectation of Treatment Scale is completed after the description of the intervention, before receiving any treatment and the Satisfaction with the Treatment Scale is completed after it is finished, assessing the patient´s satisfaction with the intervention.
Opinion Questionnaire about the intervention. | Through intervention completion, an average of 12 weeks
  It assesses participants' opinion about GROw online program, the videoconference sessions with the therapist, the blended format and de App. The questions refer to the satisfaction and usefulness of these components using a response scale from 0 to 10 and open-ended opinion questions.
Usability System Scale (SUS). | Through intervention completion, an average of 12 weeks
  This scale assesses the usability of a service or product and the acceptance by the users. It consists of 10 items with a response scale ranging from 1 (strongly disagree) to 5 (strongly agree).
Participants' adherence to the intervention; Drop-outs rates. | Through intervention completion, an average of 12 weeks
  The dropout rate of participants will be recorded through the GROw platform.
Participants' adherence to the intervention; number of sessions/modules completed. | Through intervention completion, an average of 12 weeks.
  The number of sessions/modules completed carried out will be collected by extracting data from the GROw platform.
Participants' adherence to the intervention; number of times participants enter the modules and review the contents. | Through intervention completion, an average of 12 weeks.
  The number of times participants enter the modules, how much time they spend on each one, and whether they review the content of the modules will be recorded through the GROw platform.
Intensity of pain from the loss. Daily by the Mobile App. | Every day; From the first day of treatment to the end of treatment (an avergage of 12 weeks).
  The application will record daily the intensity of pain from the loss experienced by the participant of the iGROw group, using a likert-type scale 0-10. Higher scores mean that the participant is experiencing a high intensity of pain from the loss and lower scores mean that the participant is experiencing a low intensity of pain from the loss on the day.
Intensity of the sadness. Daily by the Mobile App. | Every day; From the first day of treatment to the end of treatment (an average of 12 weeks).
  The application will record daily the intensity of the sadness experienced by the participant of the iGROw group, using a likert-type scale 0-10. Higher scores mean that the participant is experiencing a high intensity of the sadness and lower scores mean that the participant is experiencing a low intensity of the sadness on the day.
Intensity of the anxiety. Daily by the Mobile App. | Every day; From the first day of treatment to the end of treatment (an average of 12 weeks).
  The application will record daily the intensity of the anxiety experienced by the participant of the iGROw group, using a likert-type scale 0-10. Higher scores mean that the participant is experiencing a high intensity of the anxiety and lower scores mean that the participant is experiencing a low intensity of the anxiety on the day.
Motivation to continue treatment. Daily by the Mobile App. | Every day; From the first day of treatment to the end of treatment (an average of 12 weeks).
  The application will record daily the motivation to continue treatment by the participant of the iGROw group, using a likert-type scale 0-10. High scores mean that the participant is very eager to continue treatment and low scores mean that the patient is very unwilling to continue treatment on the day.
Frequency of pleasant memories with the deceased loved one. Daily by the Mobile App. | Every day; From the first day of treatment to the end of treatment (an average of 12 weeks).
  The application will record daily the frequency of pleasant memories with the deceased loved one by the participant of the iGROw group, using a likert-type scale 0-4. High scores mean that the patient has had many pleasant memories with the deceased loved one and low scores mean that the participant has had very few or no pleasant memories on the day.

CONTACTS AND LOCATIONS:
Overall Officials: Soledad Quero, Ph.D and psychology, Principal Investigator — Department of Basic, Clinical Psychology and Psychobiology, Universitat Jaume I, Castellón de la Plana, Spain.; Daniel Campos, Ph.D and psychology, Study Director — Department of Psychology and Sociology, Universidad de Zaragoza, Zaragoza, Spain.
Locations (2):
- Spain (2):
  - Universitat Jaume I, Castellon, Castellón de La Plana
  - Universitat Jaume I, Castellon, Castellón

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] WHO. (2018). ICD-11 international classification of diseases for mortality and morbidity statistics (11th revision). Retrieved from https://icd.who.int/ct11_2018/ icd11_mms/en/release#/
- [Background] Wagner B, Rosenberg N, Hofmann L, Maass U. Web-Based Bereavement Care: A Systematic Review and Meta-Analysis. Front Psychiatry. 2020 Jun 24;11:525. doi: 10.3389/fpsyt.2020.00525. eCollection 2020. PMID 32670101
- [Background] Tur C, Campos D, Suso-Ribera C, Kazlauskas E, Castilla D, Zaragoza I, Garcia-Palacios A, Quero S. An Internet-delivered Cognitive-Behavioral Therapy (iCBT) for Prolonged Grief Disorder (PGD) in adults: A multiple-baseline single-case experimental design study. Internet Interv. 2022 Jul 7;29:100558. doi: 10.1016/j.invent.2022.100558. eCollection 2022 Sep. PMID 35865996
- [Background] Tur C, Campos D, Herrero R, Mor S, Lopez-Montoyo A, Castilla D, Quero S. Internet-delivered Cognitive-Behavioral Therapy (iCBT) for Adults with Prolonged Grief Disorder (PGD): A Study Protocol for a Randomized Feasibility Trial. BMJ Open. 2021 Jul 6;11(7):e046477. doi: 10.1136/bmjopen-2020-046477. PMID 34230018
- [Background] Kessler RC, Demler O, Frank RG, Olfson M, Pincus HA, Walters EE, Wang P, Wells KB, Zaslavsky AM. Prevalence and treatment of mental disorders, 1990 to 2003. N Engl J Med. 2005 Jun 16;352(24):2515-23. doi: 10.1056/NEJMsa043266. PMID 15958807
- [Background] Kazdin AE. Addressing the treatment gap: A key challenge for extending evidence-based psychosocial interventions. Behav Res Ther. 2017 Jan;88:7-18. doi: 10.1016/j.brat.2016.06.004. PMID 28110678
- [Background] Dias N, Boring E, Johnson LA, Grossoehme DH, Murphy S, Friebert S. Developing a theoretically grounded, digital, ecological momentary intervention for parental bereavement care using the ORBIT model-Phase 1. Death Stud. 2024;48(10):1015-1024. doi: 10.1080/07481187.2021.1914239. Epub 2021 Apr 29. PMID 33913789